CLINICAL TRIAL: NCT04192994
Title: Evaluation do Early Pars Plana Vitrectomy in Acute Endophthalmitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Vinicius Campos Bergamo (Unknown); Nilva Simeren Bueno de Moraes (Unknown); Luis Filipe Nakayama (Unknown); Natasha Ferreira Santos da Cruz (Unknown); Murilo Ubukata Polizelli (Unknown)
Responsible Party: Principal Investigator, Mauricio Maia, Principal Investigator, Clinical Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: END_2019
Record Dates: First submitted 2019-11-15; First posted 2019-12-10 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Endophthalmitis
MeSH Terms: conditions — Endophthalmitis | interventions — Paracentesis

STUDY DESIGN:
Intervention Model Description: Group 1: Intravitreal Antibiotic: Group 1a: intravitreal antibiotic isolated; group 1b: intravitreal antibiotic isolated + oral moxifloxacin.
  Group 2: PPV: Group 2a: PPV + intraoperative intravitreal antibiotic ; group 2b: PPV + oral moxifloxacin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Antibiotic injection (Active Comparator): A total of 0.05 ml of vancomycin 1 mg and 0.05 ml of ceftazidime 2.25 mg will be injected with a 30-gauge needle into the vitreous cavity of the affected eyes in the randomized group, as soon as the diagnosis is confirmed.
  Interventions: Procedure: Pars Plana Vitrectomy
- Group 2: Pars Plana Vitrectomy (Active Comparator): Randomized patients will undergo PPV. Briefly, a blepharostat will be placed followed by instillation of a drop of 5% iodine-povidone over the eye. Under a surgical microscope, three 23-gauge or 25-gauge sclerotomies will be performed. Vitreous core vitrectomy will be performed, and a fluid-gas exchange with balanced saline solution (BSS) or 5,000 grams of silicone oil as a vitreous substitute. At the end of surgery, all sclerotomies will be sutured with Vicryl 7.0 and a total of 0.05 ml of vancomycin 1 mg and 0.05 ml of ceftazidime 2.25 mg will be injected into the vitreous cavity. As soon as the diagnosis is confirmed.
  Interventions: Drug: Intravitreal Antibiotic Injection

INTERVENTIONS:
Drug: Intravitreal Antibiotic Injection — Intravitreal Antibiotic Injection
  Other Names: Tap Injection
  Arms: Group 2: Pars Plana Vitrectomy
Procedure: Pars Plana Vitrectomy — Pars Plana Vitrectomy
  Other Names: PPV
  Arms: Group 1: Antibiotic injection

SUMMARY:
Our study will evaluate the efficacy of early PPV in acute endophthalmitis and attempt to prove its greater effectiveness for combating infection when compared to eyes that received only intravitreal antibiotic therapy

DETAILED DESCRIPTION:
Endophthalmitis, a severe inflammatory ocular condition with profound visual impairment that can lead to irreversible visual loss, requires immediate treatment.

The only multicenter randomized trial of different forms of acute endophthalmitis treatment was the Endophthalmitis Vitrectomy Study. The study concluded that intravitreal antibiotic injection improves visual prognosis, and pars plana vitrectomy (PPV) improves the final visual acuity (VA) when performed in patients with light perception or worse VA.

Our study will evaluate the efficacy of early PPV in acute endophthalmitis and attempt to prove its greater effectiveness for combating infection when compared to eyes that received only intravitreal antibiotic therapy.

Primary Endpoint: The final VA, ocular anatomy, retinal layer anatomy, and ERG response in the intravitreal injection group will be compared with the PPV group.

Secondary Endpoint: The final VA, eyeball anatomy, retinal layer anatomy, and ERG response in the group that underwent PPV will be compared with and without oral moxifloxacin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute endophthalmitis with a history of ocular surgical procedures and a follow-up time of less than 6 weeks will be included.

Exclusion Criteria:

* Patients with endophthalmitis lasting more than 6 weeks and no history of eye surgery will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18+
Enrollment: 25 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Best Correct Visual Acuity | 1 year
  The Final Visual acuity will be measured after 1 year
Ocular Anatomy | 1 year
  The Ocular Anatomy will be evaluated after 1 year, with axial length measured by ocular ultrasound (millimeters)
Electroretinography Response (ERG Response) | 1 year
  The ERG Response will be evaluated after 1 year, measured by Electroretinography (millivolts)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Ophthalmology - UNIFESP/Hospital São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bergamo VC, Nakayama LF, de Moraes NSB, Tavares IM, De Queiroz Campos MS, Hofling-Lima AL, Maia M. Postoperative endophthalmitis treatment with antibiotics associated or not with pars plana vitrectomy: a randomized clinical trial. Int J Retina Vitreous. 2025 Feb 18;11(1):18. doi: 10.1186/s40942-025-00640-1. PMID 39966901